CLINICAL TRIAL: NCT05632562
Title: Multiparametic Metabolic and Hypoxic PET/MRI for Disease Assessment in High Grade Glioma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R22-193; 300010076 (Other: University of Alabama at Birmingham IRB)
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma | interventions — O-(2-fluoroethyl)tyrosine; (18F)fluoroethyltyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PET imaging of system L amino acid transport with FET and hypoxia imaging with FMISO (Experimental): The participant will have a plastic peripheral intravenous (IV) catheter placed in the arm for Positron emission tomography (PET) tracer and MR contrast administration. FET O-([2-[18F]fluoroethyl)-L-tyrosine and FMISO 1H-1-(3-[18F]fluoro-2-hydroxypropyl)-2-nitroimidazole will be produced by the UAB Cyclotron PET Production Facility. PET/MRI will be performed using a GE Signa PET/MRI system in the AIF with specific imaging protocols for FET and FMISO studies. Upon completion of imaging, the peripheral IV catheter will be removed. The participant will be asked to urinate to reduce bladder dose after completion of each PET acquisition.Patients enrolled in the study will be followed clinically and with standard of care brain MRI. PFS and OS will be monitored for up to 24 months after completion of FET and FMISO PET/MRI studies.
  Interventions: Drug: O-(2-[18F]Fluoroethyl)-L-tyrosine, [18F]-FET with PET/MRI

INTERVENTIONS:
Drug: O-(2-[18F]Fluoroethyl)-L-tyrosine, [18F]-FET with PET/MRI — High grade glioma patients that are planning to undergo radiation therapy (RT) and consent to this study will have up to 3 in-person study visits. The first visit will take up to 2 hours, the second visit will take up to 3 hours, and the third visit will take up to 6 hours. After both imaging visits, there will be a phone call at 24-48 hours after imaging.After confirmation of patient eligibility and consent, the administration of FET and FMISO and related procedures will be performed in the UAB Advanced Imaging Facility (AIF) at the time of first standard of care (SOC) MRI after completion of RT (typically a 4-week interval). Patients enrolled in the study will be followed clinically and with standard of care brain MRI. PFS and OS will be monitored for up to 24 months after completion of FET and FMISO PET/MRI studies. Study participants will not undergo additional study related procedures after completion of the FET-PET/MRI and FMISO-PET/MRI studies.

SUMMARY:
This feasibility study will assess the clinical potential of a new imaging approach to detect viable high grade glioma (HGG) in pediatric and adult patients after standard of care radiation therapy (RT) with or without concurrent temozolomide (TMZ). Study participants will undergo simultaneous positron emission tomography/magnetic resonance imaging (PET/MRI) with O-([2-[F-18]fluoroethyl)-L-tyrosine (FET, amino acid transport) and 1H-1-(3-[F-18]fluoro-2-hydroxypropyl)-2-nitroimidazole (FMISO, hypoxia) at the time of standard of care imaging after completion of RT. The presence of viable tumor at this time point will be assessed on a per patient basis. Study participants will be followed clinically and with standard of care (SOC) imaging for up to 2 years after completion of PET/MRI to determine the nature of lesions seen on investigational imaging and to obtain patient outcome data. The imaging data will also be used to develop a semi-automated workflow suitable for implementation in clinical trials and standard of care PET/MRI studies.

DETAILED DESCRIPTION:
Patient recruitment

Potential participants will be identified through the UAB and Children's of Alabama (CoA) Neuro-Oncology, Neurosurgery and Radiation Oncology services. Patients seen in UAB clinics and/or discussed in multi-disciplinary neuro-oncology tumor board meetings may be approached to participate in this study. Potential participants can be enrolled from the time that the plan for standard of care therapy is selected through the time of the first standard of care of MRI after radiation therapy. Given that high grade gliomas are much more frequent in adults than children, we expect to recruit mostly adults in this study.

Confirmation of patient eligibility

The following information will be collected to confirm patient eligibility prior to the administration of FET.

1. Registering physician's name.
2. Participant's sex, race and date of birth.
3. Copy of signed consent form
4. Completed eligibility checklist that has been signed and dated by a member of the study team.
5. Copy of source documentation confirming patient eligibility.

Initial Visit

Potential participants will meet with study personnel in the appropriate neuro-oncology clinic or on the 7th floor of Jefferson Tower/Quarterback Tower. For pediatric patients under the age of consent, a parent or legal guardian will provide consent, and when possible and age appropriate, the child will provide assent. Questions will be answered, and once the participant signs informed consent, blood will be drawn to measure serum creatinine and calculate estimated GFR (eGFR). In pediatric patients, this blood draw will also be used to measure cystatin C for use in eGFR calculation. Serum creatinine and cystatin C measurements will not be required if results from previous tests within the past 4 weeks are available and meet eligibility requirements. For women with childbearing potential, a serum beta-hCG pregnancy test will be drawn along with the serum creatinine blood draw; a urine pregnancy test is acceptable to avoid a blood draw if no serum creatinine measurement is needed.

PET/MRI visits

After confirmation of patient eligibility and consent, the administration of FET and FMISO and related procedures will be performed in the UAB Advanced Imaging Facility (AIF) at the time of first SOC MRI after completion of RT (typically a 4-week interval). FET and FMISO PET/MRI studies will be performed on separate days within 2 weeks of each other, and every effort will be made to perform these studies within 1 week of each other. FET-PET/MRI will typically be performed before FMISO-PET/MRI although the order can be switched if needed from due to PET tracer production or scanner scheduling. Patients will fast for at least 4 hours prior to FET administration. No fasting or other special preparation is required for FMISO studies. Upon arrival in the AIF, the patient (and their legal medical decision maker if needed) will have an opportunity to have any remaining questions answered regarding the procedure.

The participant will have a plastic peripheral intravenous (IV) catheter placed in the arm for PET tracer and MR contrast administration. FET and FMISO will be produced by the UAB Cyclotron PET Production Facility. PET/MRI will be performed using a GE Signa PET/MRI system in the AIF with specific imaging protocols for FET and FMISO studies. Upon completion of imaging, the peripheral IV catheter will be removed. The participant will be asked to urinate to reduce bladder dose after completion of each PET acquisition. The PET data will be reconstructed using OSEM algorithms with correction for radionuclide decay, randoms and scatter according to the manufacturer's standard procedure. Attenuation correction will be performed using standard MR-based attenuation correction according to the manufacturer's recommendations.

If the PET/MRI is unexpectedly unavailable, participants can undergo brain PET imaging on a GE 710 PET/CT scanner located adjacent to the PET/MRI scanner in the AIF. The PET tracer administration and PET acquisition will be identical to the protocol described previously for PET/MRI. Attenuation correction of the PET data will be based on a low dose head CT (120 kVp, 30 mAs) for the PET/CT study. Participants undergoing PET/CT will have a separately acquired MRI study using the same MRI sequences described previously for the PET/MRI study.

FET-PET/MRI protocol

The patient will be positioned in the PET/MRI scanner prior to FET administration. FET (5 mCi, 185 MBq) will be administered IV as a bolus with dynamic acquisition of brain PET/MRI data from the time of injection through 60 min after injection. The dynamic FET-PET data will be framed according to the following schedule: 12 x 5 sec, 12 x 10 sec, 6 x 20 sec, 15 x 60 sec, and 5 min for the remainder of the study. The raw PET data will be retained for possible future reprocessing.

During FET-PET acquisition, brain MRI will be acquired simultaneously. Multiplanar, multisequence contrast-enhanced MR images will be acquired based on the standard of care adult brain tumor imaging protocol at UAB and will include dynamic contrast enhanced (DCE) and diffusion weighted (DW) sequences as well as a 3D post-contrast T1 sequence to calculate contrast enhancing volumes and 3D FLAIR sequence to calculate non-enhancing peritumoral volumes.

FMISO-PET/MRI protocol

The patient will undergo IV administration of FMISO (5 mCi, 185 MBq) in an uptake room in the AIF. At approximately 4 hours after injection, the patient will be positioned on the PET/MRI scanner. A PET scan will be acquired for 30 min, and simultaneous contrast-enhanced MRI will be acquired which may include repeat DCE and DW sequences.

Participant Follow-up

The patients and/or their legally authorized representative will be asked about any adverse events at the conclusion of each PET scan. They will also be contacted by telephone 24-48 hours after PET tracer administration to confirm that the participant is in their usual state of health and to assess for any adverse events related to the imaging study. No additional follow up to assess for adverse events will be performed unless a possible study-related adverse event is reported.

Duration of Follow Up:

Patients enrolled in the study will be followed clinically and with standard of care brain MRI. PFS and OS will be monitored for up to 24 months after completion of FET and FMISO PET/MRI studies. Relevant medical information may be accessed by study team members for correlation with imaging results including clinic notes, diagnostic imaging, histopathology and genetic tumor markers relevant to HGG classification and prognosis (e.g. MGMT promotor methylation, IDH mutation status). Study participants will not undergo additional study related procedures after completion of the FET-PET/MRI and FMISO-PET/MRI studies.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed newly diagnosed grade III or grade IV glioma treated with standard of care external beam radiation therapy (RT). For diffuse midline glioma involving the pons (diffuse intrinsic pontine glioma), histological confirmation is not required. Surgical resection of the glioma prior to RT and/or concurrent temozolomide (TMZ) with RT are allowed but not required.
2. 10 years of age or older at the time of enrollment
3. Able to undergo PET/MRI without anesthesia or sedation. Minimal sedation with an anxiolytic such as alprazolam used routinely for SOC MRI is allowed.
4. Females with childbearing potential must have a negative urine β-hCG test on the day of procedure or a serum beta-hCG test within 48 hours prior to the administration of FET or FMISO.
5. ECOG performance score of 2 or better in adults. For patients less than 16 years of age, Modified Lansky score ≥ 60.
6. Life expectancy greater than 12 weeks.

Exclusion Criteria:

1. Recurrent glioma
2. Use of bevacizumab or an investigational therapeutic drug for any indication within 3 months prior to the imaging study.
3. Pregnancy or breast feeding
4. Inability to complete PET/MRI scans.
5. Significant renal dysfunction (estimated GFR < 30 mL/min)
6. Any condition which may interfere with ability to participate in or complete all study-related activities as assessed by the study team
7. Time interval greater than 12 weeks between the completion of RT and performance of FET and FMISO PET/MRI studies.

Ages: 10 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Detection of viable glioma based on PET | Up to 24 months after completing study PET/MRI visits.
  The frequency of the detection of viable tumor by FET and/or FMISO based on prespecified standardized uptake values (SUVs) and lesion to normal brain ratios will be measured. We expect to detect viable glioma in at least 25% of patients at this time point.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No